CLINICAL TRIAL: NCT00304174
Title: Translational Research on Eating Disorders: Behavioral Assessment of Motivation to Eat
Brief Title: Motivating Factors That Play a Role in Bulimia Nervosa
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: #5049/#6178R; R21MH065024-05 (NIH); DNBBS 72-NBR (Other Grant/Funding Number: DNBBS 72-NBR)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Bulimia Nervosa; Eating Disorders
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subjects with bulimia nervosa: Participants with bulimia nervosa
  Interventions: Behavioral: Motivation to eat
- Controls between 80-120% of ideal weight: Controls without bulimia nervosa
  Interventions: Behavioral: Motivation to eat

INTERVENTIONS:
Behavioral: Motivation to eat — Participants will use a computer program to earn food (a yogurt shake) by tapping on the keyboard. More taps on the keyboard will result in a larger amount of food earned by the end of the day. Once experimentation is complete on Day 1, participants will be instructed to eat as much as they can. On Days 2 and 3, participants will be given a small serving of the yogurt shake prior to beginning the computer task. Following the computer task, they will be instructed to either eat until they are comfortable (without restricting or binging), or eat as much as they can.

SUMMARY:
This study will evaluate whether people with bulimia nervosa will binge eat in a structured laboratory setting and display behavioral patterns similar to those of individuals who are dependent on drugs.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) is a serious eating disorder that is characterized by frequent uncontrolled eating binges. These binges are often followed by compensatory behavior, including the following: self-induced vomiting; misuse of laxatives, diuretics, enemas, or other medications to induce purging; fasting; or excessive exercise. If left untreated, BN can lead to many serious health issues: tooth decay; irregular menstruation; bowel damage; constipation; heart and kidney disease; intestinal damage; puffiness, especially in the face and fingers; increased hair growth on the face and body; and mineral imbalances in the body. Similar to drug abuse disorders, food-related thinking and disordered eating behavior can interfere with other occupational and social activities, as well. This study will evaluate whether people with bulimia nervosa will binge eat in a structured laboratory setting and display behavioral patterns similar to those of individuals who are dependent on drugs.

Interested participants will first report to the study site for a screening visit, during which they will be assessed for eligibility using blood tests and an interview. Eligible participants will return to the study site on 3 additional days. Participants will be asked to refrain from eating or drinking between 10 P.M. each night before reporting to the study site and 10 A.M. the next day. Each day, participants will receive breakfast, after which they will not be allowed to eat or drink until the end of the day. Participants will then use a computer program to earn food (a yogurt shake) by tapping on the keyboard. More taps on the keyboard will result in a larger amount of food earned by the end of the day. Once experimentation is complete on Day 1, participants will be instructed to eat as much as they can. On Days 2 and 3, participants will be given a small serving of the yogurt shake prior to beginning the computer task. Following the computer task, they will be instructed to either eat until they are comfortable (without restricting or binging), or eat as much as they can. A private bathroom will be available if needed. All participants, including those who did not meet criteria for participation, will be offered treatment at the study clinic once the study is complete.

ELIGIBILITY:
Inclusion Criteria:

Participants with Bulimia Nervosa:

* Meets DSM-IV criteria for bulimia nervosa
* Duration of illness is greater than 1 year
* Self-induces vomiting
* Weighs between 80% and 120% of ideal weight
* Female

Control Group:

* Weighs between 80% and 120% of ideal weight
* Female
* Ages 18-45
* No current or past psychiatric illness
* No history of eating disorder

Exclusion Criteria:

Participants with Bulimia Nervosa:

* Significant medical illness
* Current Axis I illness other than major depression
* Severe or very severe depression
* At risk for suicide
* Currently taking medication
* History of drug or alcohol abuse within the 6 months prior to study entry
* Pregnant
* Male

Control Group:

* Significant medical illness
* Currently taking medication
* History of drug or alcohol abuse within the 6 months prior to study entry
* Pregnant
* Male
* History of any eating disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants who meet DSM-IV criteria for bulimia nervosa and control participants who weigh between 80 and 120% of ideal weight
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2005-05; Primary Completion 2014-06 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Breakpoint | Measured at Day 3
Total work performed on progressive task | Measured at Day 3

CONTACTS AND LOCATIONS:
Overall Officials: B. T. Walsh, MD, Principal Investigator — New York State Psychiatric Institute at Columbia University Medical Center
Locations (1):
- Eating Disorders Clinic, New York State Psychiatric Institute, New York, New York, United States